CLINICAL TRIAL: NCT05954182
Title: Cognitive Enhancement Intervention for Creating a Healthy L.I.F.E (Lifestyle Interventions for Epilepsy)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kayela Arrotta (Other)
Responsible Party: Sponsor-Investigator, Kayela Arrotta, Principal Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 22-1005
Record Dates: First submitted 2023-06-30; First posted 2023-07-20 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Intervention (Experimental): Participants in this group will receive weekly, live, virtual group sessions for 12 weeks
  Interventions: Behavioral: Cognitive Intervention
- Control (No Intervention): Participants in this group will NOT receive the group sessions

INTERVENTIONS:
Behavioral: Cognitive Intervention — This is a virtual, group cognitive intervention. 12 live, weekly sessions will occur during the first 3 months of the study. Groups will be made up of 5-10 participants and will be led by a neuropsychologist. These sessions will include education on the brain and cognitive function as it relates to epilepsy, as well as compensatory strategies for use in daily life. After the 12 sessions, participants will be asked to continue to practice what they learned for the next nine months until their participation ends.
  Arms: Cognitive Intervention

SUMMARY:
The goal of this clinical trial is to test if cognitive interventions in those with diagnosed epilepsy can help lessen cognitive lapses and improve overall brain health.

Participants will participate in weekly, virtual group sessions led by a neuropsychologist for 12 weeks. After the 12-week mark, participants will be asked to practice what they learned for 9 more months. Participants will be asked to complete online questionnaires at certain times during the study. Researchers will compare this intervention group to another group that did not get the intervention to see if the intervention improves brain health. Participation in each of these groups will be randomly assigned. Participation in the study will last for one year.

DETAILED DESCRIPTION:
In this prospective, controlled, randomized study, investigators aim to assess the effectiveness of a cognitive intervention in improving daily function (primary outcome) in those with epilepsy. Investigators will also seek to understand how the cognitive intervention may impact objective and subjective cognitive function, quality of life, self-efficacy, locus of control, and mood (secondary outcomes).

The study team will accomplish these objectives by comparing participants that are randomly assigned to the cognitive intervention arm (12 weekly virtual group sessions led by a neuropsychologist followed by 9 months of "self-study" in addition to their standard care) to participants randomly assigned to the control arm (continuation of their standard care during the 12 months of the study). Investigators will measure the effects of the intervention using cognitive assessments, and health and quality of life questionnaires. Investigators will also collect human biospecimens of enrolled participants to assess the biologic impact of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Potential patients will be identified if they have been, or are scheduled to be seen, either in-person or virtually for a clinical visit within the Cleveland Clinic Epilepsy Center
* Adults, aged 18-60 years old, with diagnosed epilepsy
* Subjective cognitive difficulties based on patient self-report or objective cognitive deficits as determined by neuropsychological tests
* Able to independently provide informed consent
* Fluent in English
* Reading abilities at or above 8th grade level as determined by the Wide Range Achievement Test- 4th Edition (WRAT-4), Reading subtest
* Internet access and the ability to participate in online video streaming
* No history of resective or ablative epilepsy surgery
* Willing and able to participate in cognitive intervention

Exclusion Criteria:

* Patients with a current diagnosis of non-epileptic or psychogenic seizures
* Any patient that has engaged in any form of cognitive rehabilitation/intervention within the last 6 months
* Patients currently enrolled in another interventional study for epilepsy at the time of enrollment
* Anticipated or scheduled epilepsy surgery within 6 months
* Pending litigation related to the cause of epilepsy unless litigation is related to disability application
* Undergoing intensive medical treatment for serious or life-threatening illness (e.g., chemotherapy, etc.) that, in the opinion of the investigator, would impact study participation
* Serious psychiatric condition that, in the opinion of the investigator, would interfere with participation, such as schizophrenia, active psychosis, active mania, and current suicidal ideation
* Currently pregnant or less than 6 weeks postpartum
* Significant hearing and/or vision loss that, in the opinion of the investigator would preclude them from participating in remote cognitive testing and engaging in the cognitive intervention
* Participants who require an LAR or lack capacity to consent for themselves

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Everyday Functioning | 3-12 months from the beginning of the intervention
  As assessed by the Instrumental Activities of Daily Living-Compensation (IADL-C) questionnaire - Min/Max: 27-216 (higher score means worse outcome)

SECONDARY OUTCOMES:
Change in Cognitive function | 3-12 months
  As assessed by neurocognitive testing and the Memory Assessment Clinics Scale for Epilepsy (MAC-E) questionnaire - Min/Max: 30-150 (higher score means better outcome)
Change in Quality of Life | 3-12 months
  As assessed by The Quality of Life in Epilepsy (QOLIE) questionnaire - Min/Max: 0-100 (higher score means better outcome)
Change in Stress | 3-12 months
  As assessed by The Perceived Stress Scale (PSS) questionnaire - Min/Max: 0-16 (higher score means worse outcome)
Change in Mood | 3-12 months
  As assessed by The Patient Health Questionnaire (PHQ) questionnaire - Min/Max: 0-24 (higher score means worse outcome)
Change in Mood | 3-12 months
  As assessed by The Generalized Anxiety Disorder (GAD-7) questionnaire - Min/Max: 0-21 (higher score means worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Kayela Arrotta, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Motamedi G, Meador K. Epilepsy and cognition. Epilepsy Behav. 2003 Oct;4 Suppl 2:S25-38. doi: 10.1016/j.yebeh.2003.07.004. PMID 14527481
- [Background] Baxendale S. Cognitive rehabilitation and prehabilitation in people with epilepsy. Epilepsy Behav. 2020 May;106:107027. doi: 10.1016/j.yebeh.2020.107027. Epub 2020 Mar 21. PMID 32208338
- [Background] Farina E, Raglio A, Giovagnoli AR. Cognitive rehabilitation in epilepsy: An evidence-based review. Epilepsy Res. 2015 Jan;109:210-8. doi: 10.1016/j.eplepsyres.2014.10.017. Epub 2014 Nov 6. PMID 25524861